CLINICAL TRIAL: NCT03675087
Title: Assessment of Exercise Response in Chronic Fatigue Syndrome / Myalgic Encephalomyelitis.
Status: Recruiting | Type: Observational
Sponsor: Escuela Universitaria de Fisioterapia de la Once (Other)
Collaborators: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Susana García Juez, PhD candidate. Master´s degree in physiotherapy. Postgraduate and degree lecturer of Escuela Universitaria de Fisioterapia de la ONCE. Physioterapist practice in a private clinic., Escuela Universitaria de Fisioterapia de la Once
Other Study IDs: 1
Record Dates: First submitted 2018-09-02; First posted 2018-09-18 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Fatigue Syndrome, Chronic
Keywords: Work Capacity Evaluation; Fatigue Syndrome,Chronic; Exercise Tests
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the correlation between the 6-min walking test (6MWT) with gases measurement, and the peak cardiopulmonary exercise testing (CPET) using incremental cycling with gases and workload measurement, in order to determine if the 6MWT detects impairment in exercise tolerance and if it avoids the post-exertional malaise that the peak CPET causes on decreasing levels of physical activity, in participants affected by chronic fatigue syndrome/ myalgic encephalomyelitis (CFS/ME).

Physical activity level at baseline (usual activity, the parcipant will not be given any directions) will be recorded during 7 days, 24 hours/day. Afterwards, the 6MWT will be performed. After this test, the physical activity level will be collected again during 7 days, 24 hours/day. Peak CPET will be carried out 14 days after 6MWT to make sure that the basal levels are recovered, and finally, physical activity level will be collected again during 7 days, 24 hours/day.

DETAILED DESCRIPTION:
Chronic fatigue syndrome/ myalgic encephalomyelitis presents with a significant deterioration of functional capacity, which seriously affects the quality of life. The peak or maximal incremental CPET is considered valid for the evaluation of exercise tolerance of those affected by CFS/ME, but its performance causes worsening of its symptomatology, decreasing its physical activity level after the test. It has not been verified whether the 6MWT (submaximal exercise test) with gases measurement is able to assess the exercise tolerance of those affected by SFC/EM without increasing their symptoms. So far, only the correlation between another submaximal test and a peak CPET in two different groups of participants have been analyzed and proven, which it makes necessary to check adequately whether there is a correlation by performing both tests on the same participants. In addition, it is necessary to compare the degree of worsening in physical activity level that both tests produce in participants, because they have not been objectively evaluated in any previous study. It could be useful to have a more innocuous and simple test for the assessment of exercise tolerance in CFS/ME in clinical practice, in order to evaluate the benefits of treatments like rehabilitation programs. 6MWT could respond to these characteristics because it reaches an identical value in peak VO2 than in the peak CPET in other pathologies and it generates less physical stress.

This research will be developed with the utmost respect for individual human rights, according to the postulates accepted internationally by the United Nations and the European Commission (Helsinki Act of 1964 and the Oviedo Convention of 1997) and Regulation (EU) 2016/679 of the European Parliament and the Council of April 27, 2016 on Data Protection (RGPD).

Participation in this study is entirely voluntary and does not imply any risk to health. Participants are entitled to refuse to participate or to leave the study at any time they choose.

All information will be treated confidentially. If it is decided to publish the results of the study, in these publications will not include individual data or the names of the participants, only information considered globally will be included.

This study has been approved in August 2018 by the Ethics and Research Committee of the La Paz University Hospital in Madrid (HULP Code: PI-3320).

The sample sizes were calculated in order to find the significance of the Pearson linear correlation coefficient between two variables, for a unilateral hypothesis test according to the formula: n = [Z1-α + Z1- β / ½ ln (1 + r / 1-r)]^2 + 3 and the largest has been chosen, which involve studying 22 participants.

Taking into account the data of a previous study with participants of similar characteristics, a correlation of the parameters that set up the primary outcome, peak VO2 of r = 0.7 is assumed.

An expected drop out in rate of 0.474 has been estimated from the data obtained in another related study.

Accepting an alpha risk of 0.05 and a beta risk of 0.20 in a unilateral contrast, 22 participants are required to detect a positive correlation between the variables of the exercise tests, equal to or greater than those found in the study used as reference.

This size will guarantee sufficient power to detect correlation in the purpose of the study. To guarantee this power, and since there is not enough information about the previous values, an intermediate analysis of the data, will be carried out in the middle of the study to recalculate the size of the final sample.

The incidental sampling will be carried out according to a non-probabilistic system of consecutive cases of people diagnosed with CFS/ME.

Data analysis / Statistical methods:

1. Descriptive: Descriptive analysis of all variables collected will be carried out. For quantitative data, centralization and dispersion measures will be calculated according to the distribution of each variable, such as mean, standard deviation, minimum and maximum median. The qualitative data will be described by absolute frequency and percentage. It will be checked if the variables are distributed normally by means of the Kolmogórov-Smirnov test for a single sample.
2. Correlation: A bivariate analysis will be performed to observe the association between the variables obtained in the 6MWT with gases measurement and those of the peak incremental CPET; between peak VO2 in the peak CPET and the distance achieved during the 6MWT; between peak VO2 and physical activity level at baseline and after each test; and between distance achieved in the 6MWT and physical activity level at baseline and after each test. In case of normality, the Pearson product-moment correlation coefficient will be used, and if any variable is not distributed normally, the Spearman correlation analysis will be used.
3. Linear regression: If some variables of the 6MWT are strongly correlated with the corresponding variables of the peak incremental CPET, a linear regression analysis will be performed to construct a regression equation for the prediction of the peak test performance. If necessary, a multiple linear regression analysis will be carried out to control the possible confounding variables: medication intake, time of disease evolution, quality of life, multidimensional fatigue, physical activity level at baseline, age, sex, profession, weight, height and body mass index.
4. Comparison: a comparative analysis of physical activity level at baseline and physical activity levels after each of the tests and between physical activity levels after each of the tests to compare decrease in physical activity level that generate both tests; using repeated measures ANOVA for related samples, if they meet the normal distribution or, if not, the Friedman test.

In case of drop out, the data collected will be taken into account for the analysis.

The analysis will assume a confidence level (1 - α) of 0.95 (significance level α = 0.05). The program SPSS® Statistics version 20.0 (SPSS Incorporation, Chicago, USA) will be used.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed by a medical specialist in internal medicine with experience in this disease. For this, the participant must fulfill with the diagnostic criteria of CFS/ME, following the recommended criteria for the diagnosis of 2015.
* Prior signing of the informed consent.

Exclusion Criteria:

* Present any of the diagnoses considered excluding of the CFS/ME, according to the international criteria recommended for clinical diagnosis and the selection of subjects for research:

  * Primary psychiatric disorders
  * Somatoform disorders
  * or Substance abuse
* Present any of the absolute or relative contraindications, to perform exercise tests, described in previous investigations:

  * Decompensated heart failure
  * Acute myocardial infarction (less than 3 days)
  * Syncope
  * Unstable angina
  * Cardiac arrhythmia poorly controlled
  * Endocarditis, myocarditis or acute pericarditis
  * Acute pulmonary edema
  * Moderate or severe cardiac valvular stenosis
  * Suspected dissection or dissecting aortic aneurysm
  * O2 saturation at rest less than 85%
  * Acute renal failure
  * Untreated thyrotoxicosis
  * Acute infection
  * Uncontrolled hypertension (greater than 200-120 mmHg)
  * Hypertrophic obstructive cardiomyopathy
  * High-grade atrioventricular block
  * Significant pulmonary arterial hypertension
  * Advanced or risky pregnancy
  * Significant diselectrolithmia
  * Severe symptomatic aortic stenosis
  * Severe anemia
  * Pulmonary embolism
  * Acute thrombophlebitis
  * Traumatologic, orthopedic or neurological pathology that does not allow to walk or cycling.
  * Psychic incapacity to understand the instructions of the tests.
  * Present comorbidity of Multiple Chemical Sensitivity Syndrome.
  * Have performed the peak incremental CPET in the last 3 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Fatigue Syndrome/ Myalgic Encephalomyelitis affected and derived by their specialist in internal medicine from Hospital Universitario La Paz or by the Asociación de Afectados por el Síndrome de Fatiga Crónica y el Síndrome de Sensibilidad Química Múltiple de la Comunidad de Madrid, to the Escuela Universitaria de Fisioterapia de la ONCE and to the Department of Functional Tests of the Pneumology Service of the Hospital Universitario La Paz, Madrid (Spain) from October 1st, 2018 to July 1st, 2025 and that fulfill the inclusion criteria and do not present any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2019-02-27 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean Value of the Peak VO2 in both Exercise Tests (6MWT and Peak CPET) in Milillitres/ Minute. | 3 hours one day and 2 hours another day.
  The portable spirometer Oxycon Mobile CPET from JaegerTM during 6MWT or the fixed spirometer Mijnhart Oxycon during peak CPET will be used for its measuring. Those instruments are validated. Mean and standard deviation will be calculated.

SECONDARY OUTCOMES:
Mean Age of Participants in Years. | 5 minutes.
  It will be measured with the date of birth, collected by data collection sheet. Mean and standard deviation will be calculated.
Percentage of Males and Females. | 5 minutes.
  It will be collected by data collection sheet. The percentage by gender will be calculated.
Percentage of Participants´ Professions. | 5 minutes.
  Profession is an open field, works, with or without salary. It will be collected by data collection sheet. The percentage by profession will be calculated.
Mean of Time of Evolution of the Disease in Years. | 5 minutes.
  It will be measured from the date of medical diagnosis. It will be collected by data collection sheet. Mean and standard deviation will be calculated.
Percentage of Participants with Autonomic Dysfunction. | 5 minutes.
  Options yes or not, presence of orthostatic postural tachycardias and/or alterations in the Heart Rate Variability. It will be collected by data collection sheet. Percentage of participants with or without autonomic dysfunction will be calculated.
Percentage of Medications Intake. | 10 minutes.
  The type of medications consumed is an open field. It will be collected by data collection sheet. Percentage by name of medication will be calculated.
Mean of Weight in Kilograms. | 5 minutes.
  It will be measured with the Pesperson precision scale. Range 200 grams-160 kilograms. Sensitivity 100 grams. Mean and standard deviation will be calculated.
Mean of Height in Meters. | 5 minutes.
  It will be measured with the Pesperson tape height meter, range 82-200cm. Sensitivity 1mm. Mean and standard deviation will be calculated.
Mean of Body Mass Index in Kilograms/ Meters^2. | 5 minutes.
  It is calculated by dividing the weight by the square of the height with the data obtained by the two previous outcomes. Mean and standard deviation will be calculated.
Mean of Physical Activity Level at Baseline on ActivPAL 4 Micro. | 7 days.
  The time that participant spends lying, sitting, standing or walking is measured 7 days, 24 hours/day before both exercise tests. It will be registered with the activity meter ActivPAL4 micro, which is validated as an instrument for detecting the activity and as a tool for estimating energy expenditure, and whose data are reproducible. Mean and standard deviation will be calculated.
Mean Forced Vital Capacity (FVC) on Forced Spirometry in Milillitres. | 15 minutes.
  It will be performed according to the American Thoracic Society protocol with three forced spirometries The portable spirometer Oxycon Mobile CPET from JaegerTM will be used for its measuring. Mean and standard deviation will be calculated.
Mean Forced Expiratory Volume in the First Second (FEV1) on Forced Spirometry in Milillitres. | 15 minutes.
  It will be performed according to the American Thoracic Society protocol with three forced spirometries. The portable spirometer Oxycon Mobile CPET from JaegerTM will be used for its measuring. Mean and standard deviation of FEV1 will be calculated.
Mean Tiffeneau Index (FEV1 / FVC) on Forced Spirometry in Percentage. | 15 minutes.
  It is calculated with the data provided by the two previous outcomes. Mean and standard deviation will be calculated.
Mean Change from Baseline in Medications Dosage at After Both Exercise Tests (6MWT and Peak CPET). | 10 minutes on day and 10 minutes another day.
  Open field, daily medications dosage consumed before and after both tests. It will be collected by data collection sheet. Mean and standard deviation of the differences in the dose intake by type of medication will be calculated.
Mean Change from Baseline in Quality of Life Related to Health on SF-36v2 at After Both Exercise Tests. | 20 minutes one day and 20 minutes another day.
  It is measured from 0 to 100 points by the SF-36v2 (internal consistency value α of Cronbach of 0.94). This instrument provides a profile of health status, it is usually used in studies of research in the international field in the SFC/EM and a validated version is available in Spanish. Mean and standard deviation of the differences in the total questionnaire score and in the subscales of the questionnaire will be calculated.
Mean Change from Baseline in Multidimensional Fatigue on MIF:S at After Both Exercise Tests. | 10 minutes one day and 10 minutes another day.
  It is measured from 4 to 20 points with the Multidimensional Inventory of Fatigue in Spanish (MIF: S) (internal consistency value α of Cronbach of 0.91). Mean and standard deviation of the differences will be calculated.
Mean Change from Baseline in Physical Activity Level on ActivPAL 4 Micro at After each of the Exercise Tests. | 21 days, in 3 periods of 7 days.
  The mean change in values of the time that participant spends lying, sitting, standing or walking is measured 7 days, 24 hours/day before both exercise tests and 7 days, 24 hours/day after the 6MWT and after the peak CPET. It will be registered with the activity meter ActivPAL4 micro, which is validated as an instrument for detecting the activity and as a tool for estimating energy expenditure, and whose data are reproducible.
Mean Value of the Peak VO2 Body Weight Adjusted in 6MWT and in Peak CPET in Milillitres/ Kilograms/ Minute. | 3 hours one day and 2 hours another day.
  The portable spirometer Oxycon Mobile CPET from JaegerTM during 6MWT or the fixed spirometer Mijnhart Oxycon during peak CPET will be used for its measuring. Those instruments are validated. Mean and standard deviation will be calculated.
Percentage of Exercise Tolerance. | 3 hours one day and 2 hours another day.
  Class 1, 2, 3 or 4, classification of the impairment in exercise tolerance of the American Medical Association that is based on the values of percentage of peak VO2 body weight adjusted achieved during the exercise tests in accordance with the values of overall population. Percentage of participants in each class will be calculated.
Mean Distance on the 6MWT in Metres. | 3 hours.
  It will be obtained by the 6MWT with the American Thoracic Society protocol. Mean and standard deviation will be calculated.
Mean Peak Work Load on the Peak CPET in Watts. | 2 hours.
  It is measured through the Jaeger 900 cycle ergometer during the peak CPET with Snell CR. et al protocol. Mean and standard deviation of participants´ peak work load will be calculated.
Mean Change from Baseline in O2 Saturation on Spirometer at After each of the Exercise Tests. | 3 hours one day and 2 hours another day.
  It is measured in percentage with a portable spirometer Oxycon Mobile CPET of JaegerTM in the 6MWT or with a fixed spirometer Mijnhart Oxycon in the peak CPET. Mean and standard deviation will be calculated.
Mean Change from Baseline in Heart Rate on Pulsiometer or Electrocardiogram at Maximum Hearth Rate in both Exercise Tests. | 3 hours one day and 2 hours another day.
  It is measured in beats per minute with the heart rate sensor of the Polar TM31 band in 6MWT or with the 12-lead JaegerTM ECG in the peak CPET. Mean and standard deviation will be calculated.
Mean Change from Baseline in Heart Rate on Pulsiometer or Elecrocardiogram at After each of the Exercise Tests. | 3 hours one day and 2 hours another day.
  It is measured in beats per minute with the heart rate sensor of the Polar TM31 band in the 6MWT or with the 12-lead JaegerTM ECG in the peak CPET. Mean and standard deviation of the differences in hearth rate between baseline and after the 6MWT or peak CPET will be calculated.
Mean Change from Baseline in Blood Pressure on Tensiometer at After each of the Exercise Tests. | 3 hours one day and 2 hours another day.
  It is measured in mmHg with Suntech Oscar 2 tensionmeter in the 6MWT or Riester tensionmeter in the peak CPET. Mean and standard deviation will be calculated.
Mean Change from Baseline in Total Heart Rate Variability on Pulsiometer or Electrocardiogram at After each of the Exercise Tests. | 3 hours one day and 2 hours another day.
  It will be measured in milliseconds, standard deviation of all the variations in the time interval between heartbeats measured with the heart rate sensor of the TM31 Polar band in the 6MWT or with the 12-lead JaegerTM ECG in the peak CPET. Mean and standard deviation will be calculated.
Mean of the Maximum Heart Rate in Percentage. | 3 hours one day and 2 hours another day.
  It will be calculated with the value of the maximum heart rate reached and the maximum theoretical heart rate (220-patient's age) in the 6MWT and in the peak CPET. Mean and standard deviation will be calculated.
Mean Change from Baseline in VO2 on Spirometer at the Peak VO2 of the 6MWT and the Peak CPET. | 3 hours one day and 2 hours another day.
  It is measured in millilitres/ minute with a portable spirometer Oxycon Mobile CPET of JaegerTM in the 6MWT or with a fixed spirometer Mijnhart Oxycon in the peak CPET. Mean and standard deviation will be calculated.
Mean Change from Baseline in VO2 Body Weight Adjusted on Spirometer at the Peak VO2 of both Exercise Tests. | 3 hours one day and 2 hours another day.
  It is measured in millilitres/ minute /kilograms with a portable spirometer Oxycon Mobile CPET of JaegerTM in the 6MWT or with a fixed spirometer Mijnhart Oxycon in the peak CPET. Mean and standard deviation will be calculated.
Mean Change from Baseline in Oxygen Pulse on Spirometer at the Peak VO2 of both Exercise Tests. | 3 hours one day and 2 hours another day.
  It will be measured in millilitre/ cycle with a portable spirometer Oxycon Mobile CPET of JaegerTM in the 6MWT or with a fixed spirometer Mijnhart Oxycon in the peak CPET. Mean and standard deviation in differences in oxygen pulse at baseline and at peak VO2 in both exercise tests will be calculated.
Mean Change from Baseline in CO2 Production on Spirometer at the Peak VO2 of both Exercise Tests. | 3 hours one day and 2 hours another day.
  It will be measured in millilitre/ min with a portable spirometer Oxycon Mobile CPET of JaegerTM in the 6MWT or with a fixed spirometer Mijnhart Oxycon in the peak CPET. Mean and standard deviation in differences in CO2 production between baseline and peak VO2 in both exercise tests will be calculated.
Mean Change from Baseline in Respiratory Exchange Ratio (RER) at the Peak VO2 of both Exercise Tests. | 3 hours one day and 2 hours another day.
  It will be measured in millilitres/ minute, is calculated with the values of O2 consumption and CO2 production before tests and at peak VO2 of both exercise tests. Mean and standard deviation will be calculated.
Mean Change from Baseline in Minute Ventilation at the Peak VO2 of both Exercise Tests. | 3 hours one day and 2 hours another day.
  It will be measured in litres/ minute with a portable spirometer Oxycon Mobile CPET of JaegerTM in the 6MWT or with a fixed spirometer Mijnhart Oxycon in the peak CPET. Mean and standard deviation of differences between baseline and at peak VO2 of both exercise tests will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ana B Varas-de-la-Fuente, Chair, Study Chair — Escuela Universitaria de Fisioterapia de la Once; Susana García-Juez, Principal Investigator — Escuela Universitaria de Fisioterapia de la Once
Locations (1):
- Escuela Universitaria de Fisioterapia de la ONCE, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennett RM. Fibromyalgia and chronic fatigue syndrome. In: Goldman L, Ausiello DA, eds. Cecil Medicine. 23rd ed. Philadelphia, Pa: Saunders Elsevier; 2007. Chapter 295.
- [Background] Fukuda K, Straus SE, Hickie I, Sharpe MC, Dobbins JG, Komaroff A. The chronic fatigue syndrome: a comprehensive approach to its definition and study. International Chronic Fatigue Syndrome Study Group. Ann Intern Med. 1994 Dec 15;121(12):953-9. doi: 10.7326/0003-4819-121-12-199412150-00009. PMID 7978722
- [Background] World Health Organization. International statistical classiﬁcation of diseases and related health problems. 10th revision. Fifth edition. 2016. [internet]. Ginebra: World Health Organization; 2016. In: http://apps.who.int/classifications/icd10/browse/2016/en.
- [Background] Engleberg N. Síndrome de fatiga crónica. En: Mandell GL, Bennett JE, Dolin R, editores, Douglas RG, colaborador. Mandell, Douglas, y Bennett. Enfermedades Infecciosas: principios y práctica. 5ª ed. Buenos Aires: Ed. Panamericana, 2002. p.1871-1877.
- [Background] Richardson RD, Engel CC Jr. Evaluation and management of medically unexplained physical symptoms. Neurologist. 2004 Jan;10(1):18-30. doi: 10.1097/01.nrl.0000106921.76055.24. PMID 14720312
- [Background] Johnston S, Brenu EW, Staines D, Marshall-Gradisnik S. The prevalence of chronic fatigue syndrome/ myalgic encephalomyelitis: a meta-analysis. Clin Epidemiol. 2013;5:105-10. doi: 10.2147/CLEP.S39876. Epub 2013 Mar 26. PMID 23576883
- [Background] Fernandez AA, Martin AP, Martinez MI. [Chronic fatigue syndrome. Consensus document]. Aten Primaria. 2009 Oct;41(10):529-31. doi: 10.1016/j.aprim.2009.06.013. Epub 2009 Sep 9. No abstract available. Spanish. PMID 19740570
- [Background] Baker R, Shaw EJ. Diagnosis and management of chronic fatigue syndrome or myalgic encephalomyelitis (or encephalopathy): summary of NICE guidance. BMJ. 2007 Sep 1;335(7617):446-8. doi: 10.1136/bmj.39302.509005.AE. No abstract available. PMID 17762037
- [Background] Collin SM, Crawley E, May MT, Sterne JA, Hollingworth W; UK CFS/ME National Outcomes Database. The impact of CFS/ME on employment and productivity in the UK: a cross-sectional study based on the CFS/ME national outcomes database. BMC Health Serv Res. 2011 Sep 15;11:217. doi: 10.1186/1472-6963-11-217. PMID 21923897
- [Background] Russell AS, Gulliver WP, Irvine EJ, Albani S, Dutz JP. Quality of life in patients with immune-mediated inflammatory diseases. J Rheumatol Suppl. 2011 Nov;88:7-19. doi: 10.3899/jrheum.110899. PMID 22045973
- [Background] Jason LA, Benton MC, Valentine L, Johnson A, Torres-Harding S. The economic impact of ME/CFS: individual and societal costs. Dyn Med. 2008 Apr 8;7:6. doi: 10.1186/1476-5918-7-6. PMID 18397528
- [Background] Beard DD. Chronic fatigue syndrome clinical practice guidelines: psychological factors. Med J Aust. 2002 Nov 4;177(9):526; author reply 526-7. doi: 10.5694/j.1326-5377.2002.tb04937.x. No abstract available. PMID 12465628
- [Background] Turnbull N, Shaw EJ, Baker R, Dunsdon S, Costin N, Britton G, et al. National Institute for Health and Clinical Excellence. Chronic fatigue syndrome/myalgic encephalomyelitis (or encephalopathy): diagnosis and management of CFS/ME in adults and children. London: Royal College of General Practitioners; 2007. In: http://guidance.nice.org.uk/CG053
- [Background] Nijs J, Meeus M, Van Oosterwijck J, Ickmans K, Moorkens G, Hans G, De Clerck LS. In the mind or in the brain? Scientific evidence for central sensitisation in chronic fatigue syndrome. Eur J Clin Invest. 2012 Feb;42(2):203-12. doi: 10.1111/j.1365-2362.2011.02575.x. Epub 2011 Jul 27. PMID 21793823
- [Background] Twisk FN. The status of and future research into Myalgic Encephalomyelitis and Chronic Fatigue Syndrome: the need of accurate diagnosis, objective assessment, and acknowledging biological and clinical subgroups. Front Physiol. 2014 Mar 27;5:109. doi: 10.3389/fphys.2014.00109. eCollection 2014. PMID 24734022
- [Background] Committee on the Diagnostic Criteria for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome; Board on the Health of Select Populations; Institute of Medicine. Beyond Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: Redefining an Illness. Washington (DC): National Academies Press (US); 2015 Feb 10. Available from http://www.ncbi.nlm.nih.gov/books/NBK274235/ PMID 25695122
- [Background] Sharpe M. The report of the Chief Medical Officer's CFS/ME working group: what does it say and will it help? Clin Med (Lond). 2002 Sep-Oct;2(5):427-9. doi: 10.7861/clinmedicine.2-5-427. PMID 12448589
- [Background] Carruthers BM, Jain AK, DeMeirleir KL, Peterson DL, Klimas NG, Lerner AM, et al. Myalgic Encephalomyelitis/chronic fatigue syndrome: Clinical working case definition, diagnostic and treatments protocols. Journal of Chronic Fatigue Syndrome. 2003;11:7-115.
- [Background] Jason L, Evans M, Porter N, Brown M, Brown A, Hunnell J, et al. The development of a revised Canadian myalgic encephalomyelitis chronic fatigue syndrome case definition. Am J Biochem Biotechnol. 2010;6(2):120-135
- [Background] Carruthers BM, van de Sande MI, De Meirleir KL, Klimas NG, Broderick G, Mitchell T, Staines D, Powles AC, Speight N, Vallings R, Bateman L, Baumgarten-Austrheim B, Bell DS, Carlo-Stella N, Chia J, Darragh A, Jo D, Lewis D, Light AR, Marshall-Gradisnik S, Mena I, Mikovits JA, Miwa K, Murovska M, Pall ML, Stevens S. Myalgic encephalomyelitis: International Consensus Criteria. J Intern Med. 2011 Oct;270(4):327-38. doi: 10.1111/j.1365-2796.2011.02428.x. Epub 2011 Aug 22. PMID 21777306
- [Background] Cairns R, Hotopf M. A systematic review describing the prognosis of chronic fatigue syndrome. Occup Med (Lond). 2005 Jan;55(1):20-31. doi: 10.1093/occmed/kqi013. PMID 15699087
- [Background] Pheley AM, Melby D, Schenck C, Mandel J, Peterson PK. Can we predict recovery in chronic fatigue syndrome? Minn Med. 1999 Nov;82(11):52-6. PMID 10589213
- [Background] Mulrow CD, Ramirez G, Cornell JE, Allsup K. Defining and managing chronic fatigue syndrome. Evid Rep Technol Assess (Summ). 2001 Sep;(42):1-4. No abstract available. PMID 11840862
- [Background] Rakib A, White PD, Pinching AJ, Hedge B, Newbery N, Fakhoury WK, Priebe S. Subjective quality of life in patients with chronic fatigue syndrome. Qual Life Res. 2005 Feb;14(1):11-9. doi: 10.1007/s11136-004-1693-y. PMID 15789937
- [Background] Anderson VR, Jason LA, Hlavaty LE. A qualitative natural history study of ME/CFS in the community. Health Care Women Int. 2014 Jan;35(1):3-26. doi: 10.1080/07399332.2012.684816. Epub 2013 Feb 27. PMID 23445264
- [Background] Taylor RR, O'Brien J, Kielhofner G, Lee SW, Katz B, Mears C. The occupational and quality of life consequences of chronic fatigue syndrome/myalgic encephalomyelitis in young people. Br J Occup Ther. 2010 Nov 1;73(11):524-530. doi: 10.4276/030802210X12892992239233. PMID 22102767
- [Background] Nacul LC, Lacerda EM, Campion P, Pheby D, Drachler Mde L, Leite JC, Poland F, Howe A, Fayyaz S, Molokhia M. The functional status and well being of people with myalgic encephalomyelitis/chronic fatigue syndrome and their carers. BMC Public Health. 2011 May 27;11:402. doi: 10.1186/1471-2458-11-402. PMID 21619607
- [Background] Twisk FN. Accurate diagnosis of myalgic encephalomyelitis and chronic fatigue syndrome based upon objective test methods for characteristic symptoms. World J Methodol. 2015 Jun 26;5(2):68-87. doi: 10.5662/wjm.v5.i2.68. eCollection 2015 Jun 26. PMID 26140274
- [Background] Jason LA, Sunnquist M, Brown A, Evans M, Vernon SD, Furst J, Simonis V. Examining case definition criteria for chronic fatigue syndrome and myalgic encephalomyelitis. Fatigue. 2014 Jan 1;2(1):40-56. doi: 10.1080/21641846.2013.862993. PMID 24511456
- [Background] Watz H, Waschki B, Meyer T, Magnussen H. Physical activity in patients with COPD. Eur Respir J. 2009 Feb;33(2):262-72. doi: 10.1183/09031936.00024608. Epub 2008 Nov 14. PMID 19010994
- [Background] Ryan CG, Grant PM, Tigbe WW, Granat MH. The validity and reliability of a novel activity monitor as a measure of walking. Br J Sports Med. 2006 Sep;40(9):779-84. doi: 10.1136/bjsm.2006.027276. Epub 2006 Jul 6. PMID 16825270
- [Background] Rabinovich RA, Louvaris Z, Raste Y, Langer D, Van Remoortel H, Giavedoni S, Burtin C, Regueiro EM, Vogiatzis I, Hopkinson NS, Polkey MI, Wilson FJ, Macnee W, Westerterp KR, Troosters T; PROactive Consortium. Validity of physical activity monitors during daily life in patients with COPD. Eur Respir J. 2013 Nov;42(5):1205-15. doi: 10.1183/09031936.00134312. Epub 2013 Feb 8. PMID 23397303
- [Background] American Medical Association. Guides to the evaluation of permanent impairment. 5ª ed. Chicago: American Medical Association; 2001.
- [Background] Sargent C, Scroop GC, Nemeth PM, Burnet RB, Buckley JD. Maximal oxygen uptake and lactate metabolism are normal in chronic fatigue syndrome. Med Sci Sports Exerc. 2002 Jan;34(1):51-6. doi: 10.1097/00005768-200201000-00009. PMID 11782647
- [Background] Klimas N, Patarca R. Disability and chronic fatigue syndrome: clinical, legal and patient perspectives. Binghamton NY: Haworth Medical Press; 1997.
- [Background] Ciccolella ME, Boone T, Davenport T. Part II. Legal aspects of aerobic capacity: objective evidence of the ability to work. PEPonline. 2011 septiembre; 14 (9): 11. In: https://www.asep.org/asep/asep/Part%20II%20Legal%20MARGARET%20CICCOLELLA.pdf.
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Erratum: ATS Statement: Guidelines for the Six-Minute Walk Test. Am J Respir Crit Care Med. 2016 May 15;193(10):1185. doi: 10.1164/rccm.19310erratum. No abstract available. PMID 27174486
- [Background] Strahler J, Fischer S, Nater UM, Ehlert U, Gaab J. Norepinephrine and epinephrine responses to physiological and pharmacological stimulation in chronic fatigue syndrome. Biol Psychol. 2013 Sep;94(1):160-6. doi: 10.1016/j.biopsycho.2013.06.002. Epub 2013 Jun 13. PMID 23770415
- [Background] Lewis I, Pairman J, Spickett G, Newton JL. Clinical characteristics of a novel subgroup of chronic fatigue syndrome patients with postural orthostatic tachycardia syndrome. J Intern Med. 2013 May;273(5):501-10. doi: 10.1111/joim.12022. Epub 2013 Jan 7. PMID 23206180
- [Background] Nijs J, Ickmans K. Postural orthostatic tachycardia syndrome as a clinically important subgroup of chronic fatigue syndrome: further evidence for central nervous system dysfunctioning. J Intern Med. 2013 May;273(5):498-500. doi: 10.1111/joim.12034. Epub 2013 Feb 8. No abstract available. PMID 23331489
- [Background] Meeus M, Goubert D, De Backer F, Struyf F, Hermans L, Coppieters I, De Wandele I, Da Silva H, Calders P. Heart rate variability in patients with fibromyalgia and patients with chronic fatigue syndrome: a systematic review. Semin Arthritis Rheum. 2013 Oct;43(2):279-87. doi: 10.1016/j.semarthrit.2013.03.004. Epub 2013 Jul 6. PMID 23838093
- [Background] Stewart JM, Medow MS, Messer ZR, Baugham IL, Terilli C, Ocon AJ. Postural neurocognitive and neuronal activated cerebral blood flow deficits in young chronic fatigue syndrome patients with postural tachycardia syndrome. Am J Physiol Heart Circ Physiol. 2012 Mar 1;302(5):H1185-94. doi: 10.1152/ajpheart.00994.2011. Epub 2011 Dec 16. PMID 22180650
- [Background] Vilagut G, Valderas JM, Ferrer M, Garin O, Lopez-Garcia E, Alonso J. [Interpretation of SF-36 and SF-12 questionnaires in Spain: physical and mental components]. Med Clin (Barc). 2008 May 24;130(19):726-35. doi: 10.1157/13121076. Spanish. PMID 18570798
- [Background] American Thoracic Society Committee in Proficiency Standars for Pulmonary Function Laboratories: Standarization of Spirometry- 1987 update. Am Rev Respir Dis. 1981; 136:1299-1307.
- [Background] Overstreet BS, Bassett DR Jr, Crouter SE, Rider BC, Parr BB. Portable open-circuit spirometry systems. J Sports Med Phys Fitness. 2017 Mar;57(3):227-237. doi: 10.23736/S0022-4707.16.06049-7. Epub 2016 Feb 10. PMID 26861831
- [Background] Beaver WL, Wasserman K, Whipp BJ. A new method for detecting anaerobic threshold by gas exchange. J Appl Physiol (1985). 1986 Jun;60(6):2020-7. doi: 10.1152/jappl.1986.60.6.2020. PMID 3087938
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Result] Hardt J, Buchwald D, Wilks D, Sharpe M, Nix WA, Egle UT. Health-related quality of life in patients with chronic fatigue syndrome: an international study. J Psychosom Res. 2001 Aug;51(2):431-4. doi: 10.1016/s0022-3999(01)00220-3. PMID 11516765
- [Result] VanNess JM, Stevens SR, Bateman L, Stiles TL, Snell CR. Postexertional malaise in women with chronic fatigue syndrome. J Womens Health (Larchmt). 2010 Feb;19(2):239-44. doi: 10.1089/jwh.2009.1507. PMID 20095909
- [Result] Schafer C, Evans M, Jason LA, So S, Brown A. Measuring substantial reductions in activity. J Prev Interv Community. 2015;43(1):5-19. doi: 10.1080/10852352.2014.973242. PMID 25584524
- [Result] Thorpe T, McManimen S, Gleason K, Stoothoff J, Newton JL, Strand EB, Jason LA. Assessing current functioning as a measure of significant reduction in activity level. Fatigue. 2016;4(3):175-188. doi: 10.1080/21641846.2016.1206176. Epub 2016 Jul 19. PMID 28217427
- [Result] Jason L, Brown M, Evans M, Anderson V, Lerch A, Brown A, Hunnell J, Porter N. Measuring substantial reductions in functioning in patients with chronic fatigue syndrome. Disabil Rehabil. 2011;33(7):589-98. doi: 10.3109/09638288.2010.503256. Epub 2010 Jul 9. PMID 20617920
- [Result] Davenport TE, Stevens SR, Baroni K, Van Ness JM, Snell CR. Reliability and validity of Short Form 36 Version 2 to measure health perceptions in a sub-group of individuals with fatigue. Disabil Rehabil. 2011;33(25-26):2596-604. doi: 10.3109/09638288.2011.582925. Epub 2011 Jun 20. PMID 21682669
- [Result] De Becker P, Roeykens J, Reynders M, McGregor N, De Meirleir K. Exercise capacity in chronic fatigue syndrome. Arch Intern Med. 2000 Nov 27;160(21):3270-7. doi: 10.1001/archinte.160.21.3270. PMID 11088089
- [Result] Javierre C, Alegre J, Ventura JL, García-Quintana A, Segura R, Suarez A, et al. Physiological Responses to Arm and Leg Exercise in Women Patients with Chronic Fatigue Syndrome. Journal of Chronic Fatigue Syndrome. 2007;14(1):43-53.
- [Result] Snell CR, Stevens SR, Davenport TE, Van Ness JM. Discriminative validity of metabolic and workload measurements for identifying people with chronic fatigue syndrome. Phys Ther. 2013 Nov;93(11):1484-92. doi: 10.2522/ptj.20110368. Epub 2013 Jun 27. PMID 23813081
- [Result] Keller BA, Pryor JL, Giloteaux L. Inability of myalgic encephalomyelitis/chronic fatigue syndrome patients to reproduce VO(2)peak indicates functional impairment. J Transl Med. 2014 Apr 23;12:104. doi: 10.1186/1479-5876-12-104. PMID 24755065
- [Result] Ratter J, Radlinger L, Lucas C. Several submaximal exercise tests are reliable, valid and acceptable in people with chronic pain, fibromyalgia or chronic fatigue: a systematic review. J Physiother. 2014 Sep;60(3):144-50. doi: 10.1016/j.jphys.2014.06.011. Epub 2014 Jul 30. PMID 25084634
- [Result] Fotheringham I, Meakin G, Punekar YS, Riley JH, Cockle SM, Singh SJ. Comparison of laboratory- and field-based exercise tests for COPD: a systematic review. Int J Chron Obstruct Pulmon Dis. 2015 Mar 19;10:625-43. doi: 10.2147/COPD.S70518. eCollection 2015. PMID 25834421
- [Result] Pankoff B, Overend T, Lucy D, White K. Validity and responsiveness of the 6 minute walk test for people with fibromyalgia. J Rheumatol. 2000 Nov;27(11):2666-70. PMID 11093451
- [Result] King S, Wessel J, Bhambhani Y, Maikala R, Sholter D, Maksymowych W. Validity and reliability of the 6 minute walk in persons with fibromyalgia. J Rheumatol. 1999 Oct;26(10):2233-7. PMID 10529146
- [Result] Troosters T, Vilaro J, Rabinovich R, Casas A, Barbera JA, Rodriguez-Roisin R, Roca J. Physiological responses to the 6-min walk test in patients with chronic obstructive pulmonary disease. Eur Respir J. 2002 Sep;20(3):564-9. doi: 10.1183/09031936.02.02092001. PMID 12358329
- [Result] Datta D, Normandin E, ZuWallack R. Cardiopulmonary exercise testing in the assessment of exertional dyspnea. Ann Thorac Med. 2015 Apr-Jun;10(2):77-86. doi: 10.4103/1817-1737.151438. PMID 25829957
- [Result] Nijs J, Demol S, Wallman K. Can submaximal exercise variables predict peak exercise performance in women with chronic fatigue syndrome? Arch Med Res. 2007 Apr;38(3):350-3. doi: 10.1016/j.arcmed.2006.10.009. Epub 2007 Jan 30. PMID 17350488
- [Result] Nijs J, Zwinnen K, Meeusen R, de Geus B, De Meirleir K. Comparison of two exercise testing protocols in patients with chronic fatigue syndrome. J Rehabil Res Dev. 2007;44(4):553-9. doi: 10.1682/jrrd.2006.12.0153. PMID 18247252
- [Result] Munguia-Izquierdo D, Segura-Jimenez V, Camiletti-Moiron D, Pulido-Martos M, Alvarez-Gallardo IC, Romero A, Aparicio VA, Carbonell-Baeza A, Delgado-Fernandez M. Multidimensional Fatigue Inventory: Spanish adaptation and psychometric properties for fibromyalgia patients. The Al-Andalus study. Clin Exp Rheumatol. 2012 Nov-Dec;30(6 Suppl 74):94-102. Epub 2012 Dec 14. PMID 23261007
- [Result] Make B, Jones JF. Impairment of patients with chronic fatigue syndrome. J Chronic Fatigue Syndr. 1997;3(4):43-56.

DOCUMENTS (1):
  • Informed Consent Form (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03675087/ICF_001.pdf